CLINICAL TRIAL: NCT01039207
Title: A Phase II Evaluation of AMG 102 (Rilotumumab) (NSC #750009) in the Treatment of Persistent or Recurrent Epithelial Ovarian, Fallopian Tube, or Primary Peritoneal Carcinoma
Brief Title: Rilotumumab in Treating Patients With Persistent or Recurrent Ovarian Epithelial Cancer, Fallopian Tube Cancer, or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GOG-0170P; NCI-2011-01996 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000662115; 20070612; GOG-0170P (Other: NRG Oncology); GOG-0170P (Other: CTEP); U10CA180868 (NIH); U10CA027469 (NIH)
Record Dates: First submitted 2009-12-22; First posted 2009-12-24 (Estimated); Results first posted 2017-09-07 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-08

CONDITIONS: Recurrent Fallopian Tube Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Primary Peritoneal Carcinoma
MeSH Terms: conditions — Fallopian Tube Neoplasms; Ovarian Neoplasms | interventions — rilotumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (rilotumumab) (Experimental): Patients receive rilotumumab IV over 30-60 minutes on days 1 and 14. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity. Tumor tissue and blood samples may be collected periodically for further laboratory analysis.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Rilotumumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Rilotumumab — Given IV
  Other Names: AMG 102; Anti-HGF Monoclonal Antibody AMG 102; Fully Human Anti-HGF Monoclonal Antibody AMG 102

SUMMARY:
This phase II trial studies how well rilotumumab works in treating patients with ovarian epithelial, fallopian tube, or primary peritoneal cancer that has failed to respond to other therapies (persistent) or has returned after a period of improvement (recurrent). Rilotumumab is a type of drug called a monoclonal antibody, and may interfere with the ability of tumor cells to grow and spread by targeting certain cells and blocking them from working.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To estimate the proportion of patients who survive progression-free for at least 6 months and the proportion of patients who have objective tumor response (complete or partial) in patients with persistent or recurrent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma.

SECONDARY OBJECTIVES:

I. To determine the frequency and severity of adverse events associated with treatment with AMG 102 (rilotumumab) as assessed by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE).

II. To determine the duration of progression-free survival (PFS) and overall survival (OS).

TERTIARY OBJECTIVES:

I. To explore the association between a panel of biomarkers (as assayed by immunohistochemistry and mutation analysis) and measures of response to treatment with AMG 102 (rilotumumab) and clinical outcome in archived tumor tissue.

II. To evaluate circulating pre- and post-treatment levels of hepatocyte growth factor/scatter factor and markers of angiogenesis and their association with response to treatment with AMG 102 (rilotumumab) and clinical outcome.

OUTLINE:

Patients receive rilotumumab intravenously (IV) over 30-60 minutes on days 1 and 14. Courses repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 3 months for 2 years and then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have recurrent or persistent epithelial ovarian, fallopian tube, or primary peritoneal carcinoma; histologic confirmation of the original primary tumor is required via the pathology report
* All patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be >= 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or >= 20 mm when measured by chest x-ray; lymph nodes must be >= 15 mm in short axis when measured by CT or MRI
* Patient must have at least one "target lesion" to be used to assess response on this protocol as defined by RECIST 1.1; tumors within a previously irradiated field will be designated as "non-target" lesions unless progression is documented or a biopsy is obtained to confirm persistence at least 90 days following completion of radiation therapy
* Patients must not be eligible for a higher priority Gynecologic Oncology Group (GOG) protocol, if one exists; in general, this would refer to any active GOG Phase III protocol for the same patient population
* Patients who have received one prior regimen must have a GOG performance status of 0, 1, or 2

  * Patients who have received two prior regimens must have a GOG performance status of 0 or 1
* Recovery from effects of recent surgery, radiotherapy, or chemotherapy
* Major surgical procedures must have taken place > 30 days before enrollment; minor surgical procedures must have taken place > 14 days before enrollment; central venous catheter placement is allowed at any time prior to enrollment provided the patient has recovered and any surgical would has healed
* Patients should be free of active infection requiring antibiotics (with the exception of uncomplicated urinary tract infections [UTI])
* Any hormonal therapy directed at the malignant tumor must be discontinued at least one week prior to registration
* Any other prior therapy directed at the malignant tumor, including immunologic agents, must be discontinued at least three weeks prior to registration
* Patients must have had one prior platinum-based chemotherapeutic regimen for management of primary disease containing carboplatin, cisplatin, or another organoplatinum compound; this initial treatment may have included intraperitoneal therapy, high-dose therapy, consolidation, non-cytotoxic agents or extended therapy administered after surgical or non-surgical assessment
* Patients are allowed to receive, but are not required to receive, one additional cytotoxic regimen for management of recurrent or persistent disease according to the following definition:

  * Cytotoxic regimens include any agent that targets the genetic and/or mitotic apparatus of dividing cells, resulting in dose-limiting toxicity to the bone marrow and/or gastrointestinal mucosa

    * Note: Patients on this non-cytotoxic study are allowed to have received prior cytotoxic chemotherapy for management of recurrent or persistent disease, as defined above; however, patients are encouraged to enroll on second-line non-cytotoxic studies prior to receiving additional cytotoxic therapy
* Patients who have received only one prior cytotoxic regimen (platinum-based regimen for management of primary disease), must have a platinum-free interval of less than 12 months, or have progressed during platinum-based therapy, or have persistent disease after a platinum-based therapy
* Patients must NOT have received any non-cytotoxic therapy for management of recurrent or persistent disease; patients are allowed to receive, but are not required to receive, biologic (non-cytotoxic) therapy as part of their primary treatment regimen
* Absolute neutrophil count (ANC) greater than or equal to 1,500/mcl
* Platelets greater than or equal to 100,000/mcl
* Hemoglobin >= 9 g/dL
* Creatinine less than or equal to 1.5 x institutional upper limit normal (ULN)
* Bilirubin less than or equal to 1.5 x ULN
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) less than or equal to 3 x ULN
* Alkaline phosphatase less than or equal to 2.5 x ULN
* PTT (partial thromboplastin time) =< 1.5 x ULN
* International normalized ratio (INR) =< 1.5 x ULN
* Neuropathy (sensory and motor) less than or equal to CTCAE grade 1
* Proteinuria: =< 1+ (urinalysis) or < 1 g/24 hrs (24 hour urine collection)
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must meet pre-entry requirements
* Patients of childbearing potential must have a negative serum pregnancy test prior to the study entry and be practicing an effective form of contraception

Exclusion Criteria:

* Patients who have had previous treatment with AMG 102 (rilotumumab) or other hepatocyte growth factor (HGF)/MET proto-oncogene, receptor tyrosine kinase (c-met) pathway inhibitors
* Patients with a history of other invasive malignancies, with the exception of non-melanoma skin cancer and other specific malignancies as noted, are excluded if there is any evidence of other malignancy being present within the last three years; patients are also excluded if their previous cancer treatment contraindicates this protocol therapy
* Patients who have received prior radiotherapy to any portion of the abdominal cavity or pelvis OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years are excluded; prior radiation for localized cancer of the breast, head and neck, or skin is permitted, provided that it was completed more than three years prior to registration, and the patient remains free of recurrent or metastatic disease
* Patients who have received prior chemotherapy for any abdominal or pelvic tumor OTHER THAN for the treatment of ovarian, fallopian tube, or primary peritoneal cancer within the last three years are excluded; patients may have received prior adjuvant chemotherapy for localized breast cancer, provided that it was completed more than three years prior to registration, and that the patient remains free of recurrent or metastatic disease
* Patients with a past history of primary endometrial cancer are excluded unless all of the following conditions are met: stage not greater than I-B; no more than superficial myometrial invasion, without vascular or lymphatic invasion; no poorly differentiated subtypes, including papillary serous, clear cell or other International Federation of Gynecology and Obstetrics (FIGO) grade 3 lesions
* Patients with an active bleeding diathesis or on concurrent or prior (within 7 days of enrollment) therapeutic anti-coagulation therapy with warfarin, heparin, or low molecular weight heparin; the use of low-dose warfarin (=< 2 mg orally [PO] daily) for prophylaxis against central venous catheter thrombosis is allowed
* Patients with serious intercurrent infections or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by this treatment
* Patients who are pregnant or breastfeeding
* Patients with psychiatric or other conditions rendering them incapable of participating in informed consent or the requirements of this protocol
* Patients with a serious or non-healing wound
* Patients with peripheral edema or lymphedema > grade 2
* Patients with known positive human immunodeficiency virus (HIV) or hepatitis C or chronic or active hepatitis B
* Patients with thromboembolic event or ischemic event within the past 12 months, such as deep venous thrombosis, pulmonary embolism, transient ischemic attack, cerebral infarction, or myocardial infarction

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2010-10; Primary Completion 2012-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lainie Martin, Principal Investigator — NRG Oncology
Locations (28):
- United States (28):
  - Providence Saint Joseph Medical Center/Disney Family Cancer Center, Burbank, California
  - The Hospital of Central Connecticut, New Britain, Connecticut
  - Florida Hospital Orlando, Orlando, Florida
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa-Wide Oncology Research Coalition NCORP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa/Holden Comprehensive Cancer Center, Iowa City, Iowa
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Carolinas Medical Center/Levine Cancer Institute, Charlotte, North Carolina
  - Novant Health Presbyterian Medical Center, Charlotte, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Summa Akron City Hospital/Cooper Cancer Center, Akron, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Women and Infants Hospital, Providence, Rhode Island
  - Baylor All Saints Medical Center at Fort Worth, Fort Worth, Texas
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This trial was opened to patient entry on October 10, 2010 and was closed to accrual on May 10, 2011.
Groups:
- AMG 102: AMG 102 (rilotumumab) 20 mg/kg IV q 2 weeks until disease progression or adverse effects prohibit further therapy (cycle = 28 days)
Period: Overall Study
Arm/Group | AMG 102
Started | 31
Completed (Eligible and treated patients.) | 31
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Eligible and treated patients.
Arm/Group | AMG 102
Number analyzed (Participants) | 31
Age, Customized [Number; unit: participants]
  40-49 years | 4
  50-59 years | 6
  60-69 years | 9
  70-79 years | 10
  80-89 years | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 27
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Patients With Objective Tumor Response Rate (Complete Response [CR] or Partial Response [PR]) Using RECIST Version 1.1
Description: Complete and Partial Tumor Response by RECIST 1.1. RECIST 1.1 defines complete response as the disappearance of all target lesions. Any pathological lymph nodes (whether target or non-target) must have reduction in short axis to <10 mm and the disappearance of all non-target lesions and normalization of tumor marker level. Partial response is defined as at least a 30% decrease in the sum of the diameters of target lesions, taking as reference the baseline sum diameters. Only those patients who have measurable disease present at baseline, have received at least one cycle of therapy, and have had their disease re-evaluated will be considered evaluable for response. These patients will have their response classified according to the definitions stated above. Complete and partial responses are included in the objective tumor response rate.
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle during treatment then every 3 months thereafter until disease progression is confirmed; also repeat at any time if clinically indicated up to 5 years.
Population: Eligible and treated patients.
Measure: Number; unit: participants
Arm/Group | AMG 102
Number analyzed (Participants) | 31
participants
  Partial response | 0
  Complete response | 1

2. Primary Outcome: Progression-free Survival > 6 Months Using RECIST 1.0
Description: Progression-free survival (PFS) was defined as the period from study entry until disease progression, death, or the last date of contact. Progression was based on RECIST 1.1. RECIST 1.1 defines progressive disease as at least a 20% increase in the sum of the diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm. The appearance of one or more new lesions or unequivocal progression of non-target lesions is also considered progression.
Time Frame: CT scan or MRI if used to follow lesion for measurable disease every other cycle during treatment then every 3 months thereafter until disease progression is confirmed; up to 6 months.
Population: Eligible and treated patients
Measure: Number; unit: participants
Arm/Group | AMG 102
Number analyzed (Participants) | 31
participants
  Patient with PFS>6 Months | 2
  Patients with PFS<6 months | 29

3. Secondary Outcome: Incidence of Adverse Effects (Grade 3 or Higher) as Assessed by Common Terminology Criteria for Adverse Events Version 4.0
Description: Number of participants with a maximum grade of 3 or higher during the treatment period.
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment
Population: Eligible and treated patients.
Measure: Number; unit: participants
Arm/Group | AMG 102
Number analyzed (Participants) | 31
participants
  Leukopenia | 1
  Neutropenia | 1
  Cardiac | 1
  Nausea | 2
  Vomiting | 4
  Other Gastrointestinal | 7
  General and administration site | 4
  Hepatobiliary | 1
  Infections/infestations | 2
  Metabolism/nutrition | 5
  Respiratory/thoracic/mediastinal | 1
  Skin/subcutaneous | 1
  Vascular disorders | 2

4. Secondary Outcome: Duration of Overall Survival (OS)
Description: Overall survival is defined as the duration of time from study entry to time of death or the date of last contact.
Time Frame: Every cycle during treatment, then every 3 months for the first 2 years, then every six months for the next three years and then annually for the next 5 years.
Population: Eligible and treated patients. Measure type = The first quartile of the distribution since follow-up time is insufficient to obtain adequate median estimates.
Measure: Number (90% Confidence Interval); unit: months
Arm/Group | AMG 102
Number analyzed (Participants) | 31
months | 4.3 [1.9 to 5.8]

5. Secondary Outcome: Duration of Progression-free Survival (PFS)
Description: as for outcome 2
Time Frame: as for outcome 1
Population: Eligible and treated patients
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | AMG 102
Number analyzed (Participants) | 31
months | 1.8 [1.7 to 1.9]

6. Other Pre Specified Outcome: Biomarker Panel From Tumor Tissue
Description: A panel of biomarkers from fixed and embedded tumor tissue will be tested for association with measures of response to treatment including PFS and OS.
Time Frame: Baseline
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Circulating Levels of HGF/Scatter Factor (SF)
Description: Exploratory analyses will be conducted to assess the possible effects of the study regimen on the biomarkers of interest as well as associations between the biomarkers and clinical outcome (such as PFS and OS).
Time Frame: Up to 1 day prior to course 2
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Circulating Levels of Markers of Angiogenesis
Description: as for outcome 7
Time Frame: Up to 1 day prior to course 2
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment, and up to 5 years in follow-up
Arm/Group | AMG 102
All-Cause Mortality (participants affected / at risk) | 14/31
Serious Adverse Events (participants affected / at risk) | 14/31
Other Adverse Events (participants affected / at risk) | 31/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 102 (N=31)
Diarrhea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 3
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 3
Gastrointestinal Disorders - Other (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Death Nos (General disorders) | 3
Fall (Injury, poisoning and procedural complications) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 2
Thromboembolic Event (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 102 (N=31)
Anemia (Blood and lymphatic system disorders) | 20
Atrial Fibrillation (Cardiac disorders) | 1
Ventricular Tachycardia (Cardiac disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Eye Disorders - Other (Eye disorders) | 1
Blurred Vision (Eye disorders) | 2
Duodenal Obstruction (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 8
Diarrhea (Gastrointestinal disorders) | 6
Vomiting (Gastrointestinal disorders) | 11
Bloating (Gastrointestinal disorders) | 1
Small Intestinal Obstruction (Gastrointestinal disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 6
Obstruction Gastric (Gastrointestinal disorders) | 1
Mucositis Oral (Gastrointestinal disorders) | 1
Abdominal Distension (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 14
Ascites (Gastrointestinal disorders) | 2
Pain (General disorders) | 5
Localized Edema (General disorders) | 1
Edema Trunk (General disorders) | 1
Edema Limbs (General disorders) | 7
Fatigue (General disorders) | 19
Fever (General disorders) | 5
Hepatobiliary Disorders - Other (Hepatobiliary disorders) | 1
Infections And Infestations - Other (Infections and infestations) | 1
Skin Infection (Infections and infestations) | 1
Sinusitis (Infections and infestations) | 1
Peritoneal Infection (Infections and infestations) | 1
Lung Infection (Infections and infestations) | 1
Catheter Related Infection (Infections and infestations) | 1
Wound Complication (Injury, poisoning and procedural complications) | 1
Weight Loss (Investigations) | 1
Platelet Count Decreased (Investigations) | 4
Inr Increased (Investigations) | 2
Creatinine Increased (Investigations) | 2
Neutrophil Count Decreased (Investigations) | 1
Blood Bilirubin Increased (Investigations) | 2
White Blood Cell Decreased (Investigations) | 5
Aspartate Aminotransferase Increased (Investigations) | 1
Alkaline Phosphatase Increased (Investigations) | 3
Alanine Aminotransferase Increased (Investigations) | 4
Activated Partial Thromboplastin Time Prolonged (Investigations) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 3
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypomagnesemia (Metabolism and nutrition disorders) | 8
Hypokalemia (Metabolism and nutrition disorders) | 5
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Hypernatremia (Metabolism and nutrition disorders) | 1
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Anorexia (Metabolism and nutrition disorders) | 8
Pain In Extremity (Musculoskeletal and connective tissue disorders) | 3
Myalgia (Musculoskeletal and connective tissue disorders) | 2
Generalized Muscle Weakness (Musculoskeletal and connective tissue disorders) | 1
Buttock Pain (Musculoskeletal and connective tissue disorders) | 1
Back Pain (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Peripheral Sensory Neuropathy (Nervous system disorders) | 8
Peripheral Motor Neuropathy (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Memory Impairment (Nervous system disorders) | 1
Headache (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 2
Depression (Psychiatric disorders) | 2
Confusion (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 1
Urinary Incontinence (Renal and urinary disorders) | 1
Urinary Tract Pain (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 2
Reproductive System And Breast Disorders - Other (Reproductive system and breast disorders) | 1
Pelvic Pain (Reproductive system and breast disorders) | 1
Pleural Effusion (Respiratory, thoracic and mediastinal disorders) | 3
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Skin And Subcutaneous Tissue Disorders - Other (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Rash Maculo-Papular (Skin and subcutaneous tissue disorders) | 1
Nail Ridging (Skin and subcutaneous tissue disorders) | 1
Nail Loss (Skin and subcutaneous tissue disorders) | 1
Nail Discoloration (Skin and subcutaneous tissue disorders) | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2
Lymphedema (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less